CLINICAL TRIAL: NCT02783144
Title: Dexamethasone Added to Levobupivacaine in Ultrasound-guided Tranversus Abdominis Plain Block Increased the Duration of Postoperative Analgesia After Laparoscopic Cholecystectomy
Brief Title: Dexamethasone Added in Ultrasound-guided Transversus Abdominis Plain Block for Postoperative Analgesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Doctor, San Salvatore Hospital of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0024575/16
Record Dates: First submitted 2016-05-11; First posted 2016-05-26 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain
Keywords: Analgesia; Dexamethasone; Levobupivacaine; Ultrasound-guided; Tranversus Abdominis
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAP Block and Dexamethasone (Experimental): After general anesthesia and before the beginning of surgery, 4 mg of Dexamethasone are added to 20 ml of 0,375% Levobupivacaine in Ultrasound-guided Tranversus Abdominis Plain Block.
  Interventions: Procedure: TAP Block and Dexamethasone
- TAP Block and Saline (Placebo Comparator): After general anesthesia and before the beginning of surgery, 2 ml of saline are added to 20 ml of 0.375% Levobupivacaine in Ultrasound-guided Tranversus Abdominis Plain Block.
  Interventions: Other: TAP Block and saline
- TAP Block and Dexamethasone i.v. (Active Comparator): After general anesthesia and before the beginning of surgery, 20 ml of 0,375% Levobupivacaine are used in Ultrasound-guided Tranversus Abdominis Plain Block. In this group 4 mg of dexamethasone are injected intravenously.
  Interventions: Drug: TAP Block and Dexamethasone i.v.

INTERVENTIONS:
Procedure: TAP Block and Dexamethasone — After general anesthesia and before the beginning of surgery, the ultrasound-guided is performed between the internal oblique muscle and the transversus abdominis muscle and dexamethasone is added to levopubivacaine
  Other Names: TAP-Block under ultrasound guidance and dexamethasone
  Arms: TAP Block and Dexamethasone
Other: TAP Block and saline — After general anesthesia and before the beginning of surgery, the ultrasound-guided is performed between the internal oblique muscle and the transversus abdominis muscle and saline is added to levopubivacaine
  Other Names: TAP-Block under ultrasound guidance and saline
  Arms: TAP Block and Saline
Drug: TAP Block and Dexamethasone i.v. — After general anesthesia and before the beginning of surgery, the ultrasound-guided is performed between the internal oblique muscle and the transversus abdominis muscle and dexamethasone is injected intravenously
  Other Names: TAP-Block under ultrasound guidance and i.v. dexamethasone
  Arms: TAP Block and Dexamethasone i.v.

SUMMARY:
Dexamethasone Added to Levobupivacaine in Ultrasound-guided Tranversus Abdominis Plain Block Increased the Duration of Postoperative Analgesia After Laparoscopic Cholecystectomy.

DETAILED DESCRIPTION:
In the ultrasound-guided TAP-Block with Dexamethasone group, dexamethasone is added to Levobupivacaine in Ultrasound-guided Tranversus Abdominis Plain Block after Laparoscopic Cholecystectomy. In the ultrasound-guided TAP-Block with saline group, saline is added to Levobupivacaine in Ultrasound-guided Tranversus Abdominis Plain Block , after Laparoscopic Cholecystectomy. In the ultrasound-guided TAP-Block with intravenously dexamethasone group, dexamethasone is intravenously injected , after Laparoscopic Cholecystectomy. After surgery the extension of postoperative analgesia, incident and rest pain were evaluate in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA score I and II
* age 18 years

Exclusion Criteria:

* Allergy to local anesthetics
* Allergy to general anesthetics
* Allergy or intolerance to acetaminophen
* Severe renal impairment
* Severe hepatic impairment
* Congestive heart failure
* Coagulation disorders
* hypoprotidemia
* Diabetes mellitus History
* Age greater than 70 years
* Age below 18 years
* ASA Physical than 3 Status
* Lack of informed consent
* Patients unable to discernment
* Intolerance to opiates
* Peptic Ulcer
* Abuse of alcohol and / or drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Extension of analgesia, assessed in minutes after TAP block | 24 hours after surgery
  After surgery, the extension of analgesia is evaluated in minutes after TAP Block, in the first 24 hours, from operating theatre discharge.

SECONDARY OUTCOMES:
Rest pain, assessed with Visual Analog Scale | 24 hours after surgery
  Rest pain was assessed using Visual Analog Scale (10 steps scale, from 0 as no pain to 10 as the worst imaginable pain).
Incident pain, assessed with Visual Analog Scale | 24 hours after surgery
  Incident pain was assessed using Visual Analog Scale (10 steps scale, from 0 as no pain to 10 as the worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Petrucci, Principal Investigator — San Salvatore Academic Hospital of L'Aquila
Locations (1):
- Emiliano Petrucci, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No